CLINICAL TRIAL: NCT02930265
Title: Chinese People's Liberation Army General Hospital
Brief Title: Clinical Study of Liraglutide in Improving Cardiac Function for Patients With Ischemic Cardiomyopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Qian geng, Associate attending doctor, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: qs20160920
Record Dates: First submitted 2016-09-23; First posted 2016-10-12 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Ischemic Cardiomyopathy
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liraglutide intervention group (Active Comparator): Liraglutide intervention group will accept ischemic cardiomyopathy conventional drugs and Liraglutide (Novo Nordisk, specifications: 18mg / 3ml; 1.8mg subcutaneous injection of 1 / day)
  Interventions: Drug: Liraglutide
- Control group (No Intervention): Control group will accept ischemic cardiomyopathy conventional drugs and a placebo

INTERVENTIONS:
Drug: Liraglutide — Liraglutide intervention group will accept liraglutide (Novo Nordisk, specifications: 18mg / 3ml; 1.8mg subcutaneous injection of 1 / day)
  Other Names: Saxenda
  Arms: Liraglutide intervention group

SUMMARY:
It has been known that liraglutide reduces infarct size, improved left ventricular function, reduce myocardial stunning, and play a protective role in myocardial ischemia-reperfusion injury for patients with acute myocardial infarction. But it is not sure whether liraglutide can benefit patients with ischemic cardiomyopathy. This study aim to explore the effect of Liraglutide in improving cardiac function for patients with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
Investigators will enroll 400 patients with ischemic cardiomyopathy who were admitted to the Chinese PLA General Hospital. All patients enrolled in this study will collect detailed baseline clinical data, including blood, enzymes (troponin, creatine kinase), blood sugar, serum creatinine, blood lipid levels (LDL lipoprotein cholesterol, high density lipoprotein cholesterol, triglycerides, total cholesterol), brain natriuretic peptide (BNP), inflammatory markers (high sensitivity C- reactive protein, interleukin-6), endothelin (ET-1), pancreas glucagon-like peptide -1 (GLP-1) and superoxide dismutase (SOD).

The investigators randomly assign eligible patients in a 1:1 ratio to either liraglutide intervention group (N = 200) or control group (N = 200), liraglutide intervention group will accept ischemic cardiomyopathy conventional drugs and liraglutide (Novo Nordisk, specifications: 18mg / 3ml; 1.8mg subcutaneous injection of 1 / day), Control group will accept ischemic cardiomyopathy conventional drugs and a placebo.

Primary end point of the study is main adverse cardiovascular events including Recurrent myocardial infarction, recurrent angina, revascularization, all-cause death, nonfatal myocardial infarction, nonfatal stroke, hospitalization for heart failure again. Secondary end point of the study was 1) New York Heart Association functional class, 2) left ventricular ejection fraction, 3) 6-minute walk test, 4) KCCQ clinical total score, 5) changes in blood glucose levels during follow-up, blood lipid levels and body weight

ELIGIBILITY:
Inclusion Criteria:

* Patients With Ischemic Cardiomyopathy: The clinical manifestations of heart failure (NYHA class II-IV grade), evidence of cardiac dysfunction (LVEF ≤40%, and LVEDD ≥55mm) and previous coronary angiography showed one or more severe coronary artery stenosis.

Exclusion Criteria:

* Valvular heart disease
* dilated cardiomyopathy
* patients requiring emergency PCI
* patients with cardiogenic shock;
* there have been recent acute myocardial infarction in one month;
* there have been recent acute stroke in one month;
* estimated glomerular filtration over rate eGFR <30ml / min / 1.73m2 (according to MDRD formula);
* malignant tumor
* severe liver failure
* respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
main adverse cardiovascular events | Followed up for 6 months after enrolled in the study
  Primary end point of the study is main adverse cardiovascular events including Recurrent myocardial infarction, recurrent angina, revascularization, all-cause death, nonfatal myocardial infarction, nonfatal stroke, hospitalization for heart failure again

SECONDARY OUTCOMES:
New York Heart Association functional class | Followed up for 6 months after enrolled in the study
left ventricular ejection fraction | Followed up for 6 months after enrolled in the study
6-minute walk test | Followed up for 6 months after enrolled in the study
KCCQ (Kansas City cardiomyopathy questionnaire) clinical total score | Followed up for 6 months after enrolled in the study

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese People's Liberation Army General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matsubara M, Kanemoto S, Leshnower BG, Albone EF, Hinmon R, Plappert T, Gorman JH 3rd, Gorman RC. Single dose GLP-1-Tf ameliorates myocardial ischemia/reperfusion injury. J Surg Res. 2011 Jan;165(1):38-45. doi: 10.1016/j.jss.2009.03.016. Epub 2009 Apr 16. PMID 19552923
- [Background] Timmers L, Henriques JP, de Kleijn DP, Devries JH, Kemperman H, Steendijk P, Verlaan CW, Kerver M, Piek JJ, Doevendans PA, Pasterkamp G, Hoefer IE. Exenatide reduces infarct size and improves cardiac function in a porcine model of ischemia and reperfusion injury. J Am Coll Cardiol. 2009 Feb 10;53(6):501-10. doi: 10.1016/j.jacc.2008.10.033. PMID 19195607
- [Background] Noyan-Ashraf MH, Momen MA, Ban K, Sadi AM, Zhou YQ, Riazi AM, Baggio LL, Henkelman RM, Husain M, Drucker DJ. GLP-1R agonist liraglutide activates cytoprotective pathways and improves outcomes after experimental myocardial infarction in mice. Diabetes. 2009 Apr;58(4):975-83. doi: 10.2337/db08-1193. Epub 2009 Jan 16. PMID 19151200
- [Background] Marso SP, Daniels GH, Brown-Frandsen K, Kristensen P, Mann JF, Nauck MA, Nissen SE, Pocock S, Poulter NR, Ravn LS, Steinberg WM, Stockner M, Zinman B, Bergenstal RM, Buse JB; LEADER Steering Committee; LEADER Trial Investigators. Liraglutide and Cardiovascular Outcomes in Type 2 Diabetes. N Engl J Med. 2016 Jul 28;375(4):311-22. doi: 10.1056/NEJMoa1603827. Epub 2016 Jun 13. PMID 27295427
- [Background] Gejl M, Sondergaard HM, Stecher C, Bibby BM, Moller N, Botker HE, Hansen SB, Gjedde A, Rungby J, Brock B. Exenatide alters myocardial glucose transport and uptake depending on insulin resistance and increases myocardial blood flow in patients with type 2 diabetes. J Clin Endocrinol Metab. 2012 Jul;97(7):E1165-9. doi: 10.1210/jc.2011-3456. Epub 2012 Apr 27. PMID 22544917
- [Background] Lonborg J, Vejlstrup N, Kelbaek H, Botker HE, Kim WY, Mathiasen AB, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Thuesen L, Krusell LR, Jensen JS, Kober L, Treiman M, Holst JJ, Engstrom T. Exenatide reduces reperfusion injury in patients with ST-segment elevation myocardial infarction. Eur Heart J. 2012 Jun;33(12):1491-9. doi: 10.1093/eurheartj/ehr309. Epub 2011 Sep 14. PMID 21920963
- [Background] Chen WR, Tian F, Chen YD, Wang J, Yang JJ, Wang ZF, Da Wang J, Ning QX. Effects of liraglutide on no-reflow in patients with acute ST-segment elevation myocardial infarction. Int J Cardiol. 2016 Apr 1;208:109-14. doi: 10.1016/j.ijcard.2015.12.009. Epub 2015 Dec 15. PMID 26849684
- [Background] Chen WR, Shen XQ, Zhang Y, Chen YD, Hu SY, Qian G, Wang J, Yang JJ, Wang ZF, Tian F. Effects of liraglutide on left ventricular function in patients with non-ST-segment elevation myocardial infarction. Endocrine. 2016 Jun;52(3):516-26. doi: 10.1007/s12020-015-0798-0. Epub 2015 Nov 16. PMID 26573925
- [Background] Chen WR, Hu SY, Chen YD, Zhang Y, Qian G, Wang J, Yang JJ, Wang ZF, Tian F, Ning QX. Effects of liraglutide on left ventricular function in patients with ST-segment elevation myocardial infarction undergoing primary percutaneous coronary intervention. Am Heart J. 2015 Nov;170(5):845-54. doi: 10.1016/j.ahj.2015.07.014. Epub 2015 Jul 26. PMID 26542491
- [Background] Read PA, Hoole SP, White PA, Khan FZ, O'Sullivan M, West NE, Dutka DP. A pilot study to assess whether glucagon-like peptide-1 protects the heart from ischemic dysfunction and attenuates stunning after coronary balloon occlusion in humans. Circ Cardiovasc Interv. 2011 Jun;4(3):266-72. doi: 10.1161/CIRCINTERVENTIONS.110.960476. Epub 2011 May 17. PMID 21586690
- [Background] Garber A, Henry R, Ratner R, Garcia-Hernandez PA, Rodriguez-Pattzi H, Olvera-Alvarez I, Hale PM, Zdravkovic M, Bode B; LEAD-3 (Mono) Study Group. Liraglutide versus glimepiride monotherapy for type 2 diabetes (LEAD-3 Mono): a randomised, 52-week, phase III, double-blind, parallel-treatment trial. Lancet. 2009 Feb 7;373(9662):473-81. doi: 10.1016/S0140-6736(08)61246-5. Epub 2008 Sep 24. PMID 18819705
- [Background] Nauck M, Frid A, Hermansen K, Shah NS, Tankova T, Mitha IH, Zdravkovic M, During M, Matthews DR; LEAD-2 Study Group. Efficacy and safety comparison of liraglutide, glimepiride, and placebo, all in combination with metformin, in type 2 diabetes: the LEAD (liraglutide effect and action in diabetes)-2 study. Diabetes Care. 2009 Jan;32(1):84-90. doi: 10.2337/dc08-1355. Epub 2008 Oct 17. PMID 18931095
- [Background] Zinman B, Gerich J, Buse JB, Lewin A, Schwartz S, Raskin P, Hale PM, Zdravkovic M, Blonde L; LEAD-4 Study Investigators. Efficacy and safety of the human glucagon-like peptide-1 analog liraglutide in combination with metformin and thiazolidinedione in patients with type 2 diabetes (LEAD-4 Met+TZD). Diabetes Care. 2009 Jul;32(7):1224-30. doi: 10.2337/dc08-2124. Epub 2009 Mar 16. PMID 19289857
- [Background] Kim SH, Abbasi F, Lamendola C, Liu A, Ariel D, Schaaf P, Grove K, Tomasso V, Ochoa H, Liu YV, Chen YD, Reaven G. Benefits of liraglutide treatment in overweight and obese older individuals with prediabetes. Diabetes Care. 2013 Oct;36(10):3276-82. doi: 10.2337/dc13-0354. Epub 2013 Jul 8. PMID 23835684
- [Background] Zhang Y, Zhou H, Wu W, Shi C, Hu S, Yin T, Ma Q, Han T, Zhang Y, Tian F, Chen Y. Liraglutide protects cardiac microvascular endothelial cells against hypoxia/reoxygenation injury through the suppression of the SR-Ca(2+)-XO-ROS axis via activation of the GLP-1R/PI3K/Akt/survivin pathways. Free Radic Biol Med. 2016 Jun;95:278-92. doi: 10.1016/j.freeradbiomed.2016.03.035. Epub 2016 Mar 31. PMID 27038735